CLINICAL TRIAL: NCT05559983
Title: A Phase I, Multicenter, Observer-Blinded, Randomized, Placebo-Controlled, Dose Escalation Trial to Evaluate the Safety and Immunogenicity of the OSP:rTTHc Cholera Conjugate Vaccine in 19 to 45 Years Old Healthy Korean Participants
Brief Title: Dose Escalation Study to Evaluate the Safety and Immunogenicity of the Cholera Conjugate Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: EuBiologics Co.,Ltd (Industry); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVI-CCV-001
Record Dates: First submitted 2022-09-21; First posted 2022-09-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cholera Vaccination Reaction
Keywords: Cholera Conjugate Vaccine; O Specific Polysaccharide; Recombinant Tetanus Toxoid Heavy Chain Fragment

STUDY DESIGN:
Intervention Model Description: The first fifty participant in the study will be enrolled into cohort A and receive low antigen product with or without adjuvant, or placebo. The Safety Monitoring Committee (SMC) and the independent Data Safety Monitoring Board (DSMB) will review the safety data collected through seven days after the second dose vaccination of the cohort A before the study enrollment can progress to cohort B (middle dose). Dose escalation to cohort C (high dose) will follow the same procedures.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study investigators, study nurse, and those assessing clinical outcomes, and laboratory analysis will be blinded to investigational product allocation until database lock for the final analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OSP:rTTHc Cholera Conjugate Vaccine (Experimental): 2 doses @0.5 mL of test vaccine administered intramuscularly in deltoid region at 4 weeks apart
  Interventions: Biological: OSP:rTTHc Cholera Conjugate Vaccine Cohort A; Biological: OSP:rTTHc Cholera Conjugate Vaccine Cohort B; Biological: OSP:rTTHc Cholera Conjugate Vaccine Cohort C
- OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate adjuvant (Experimental): 2 doses @0.5 mL of test vaccine administered intramuscularly in deltoid region at 4 weeks apart
  Interventions: Biological: OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate adjuvant Cohort A; Biological: OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate adjuvant Cohort B; Biological: OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate adjuvant Cohort C
- Placebo (Placebo Comparator): 2 doses @0.5 mL of Sterile 0.9% sodium chloride administered intramuscularly in deltoid region at 4 weeks apart
  Interventions: Other: Placebo Cohort A; Other: Placebo Cohort B; Other: Placebo Cohort C

INTERVENTIONS:
Biological: OSP:rTTHc Cholera Conjugate Vaccine Cohort A — OSP:rTTHc Cholera Conjugate Vaccine without Aluminum phosphate with dose formulation 5 µg of OSP:rTTHc
  Arms: OSP:rTTHc Cholera Conjugate Vaccine
Biological: OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate adjuvant Cohort A — OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate with dose formulation 5 µg of OSP:rTTHc
  Arms: OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate adjuvant
Other: Placebo Cohort A — Sterile 0.9% sodium chloride
  Arms: Placebo
Biological: OSP:rTTHc Cholera Conjugate Vaccine Cohort B — OSP:rTTHc Cholera Conjugate Vaccine without Aluminum phosphate with dose formulation 10 µg of OSP:rTTHc
  Arms: OSP:rTTHc Cholera Conjugate Vaccine
Biological: OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate adjuvant Cohort B — OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate with dose formulation 10 µg of OSP:rTTHc
  Arms: OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate adjuvant
Other: Placebo Cohort B — Sterile 0.9% sodium chloride
  Arms: Placebo
Biological: OSP:rTTHc Cholera Conjugate Vaccine Cohort C — OSP:rTTHc Cholera Conjugate Vaccine without Aluminum phosphate with dose formulation 25 µg of OSP:rTTHc
  Arms: OSP:rTTHc Cholera Conjugate Vaccine
Biological: OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate adjuvant Cohort C — OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate with dose formulation 25 µg of OSP:rTTHc
  Arms: OSP:rTTHc Cholera Conjugate Vaccine with Aluminum phosphate adjuvant
Other: Placebo Cohort C — Sterile 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
This Phase I, first-in-human study is intended to primarily determine the safety of the dose range with or without Aluminum phosphate adjuvant expected to be needed for later clinical studies, to determine the nature of adverse reactions (i.e., safety profile) and to secondly assess the Aluminum phosphate humoral immune responses in non-endemic population to guide future dose selection.

DETAILED DESCRIPTION:
A total of 150 eligible participants will be recruited in 3 sequential dose cohorts: low-dose 5 µg, medium-dose 10 µg, and high-dose 25 µg. In each dose cohorts, the participants will be randomized in a blinded manner into three arms (vaccine antigen with aluminum phosphate, vaccine antigen without Aluminum phosphate or placebo) in 2:2:1 ratio. All the participants will receive two intramuscular injections of 0.5 mL of the designated study vaccine or placebo on deltoid muscle, on Days 0 and 28.

The DSMB will review the safety data and approve dose escalation before investigational product injection of the next cohort is initiated.

The study primary objective is to evaluate the safety of the O Specific Polysaccharide recombinant Tetanus Toxoid Heavy Chain Fragment (OSP:rTTHc) cholera conjugate vaccine (CCV) after each dose vaccination.

The secondary objectives are:

* To evaluate the Antibody response to OSP IgG against V. cholerae O1 after each dose vaccination of OSP:rTTHc CCV/placebo compared to pre-vaccination.
* To evaluate the serum vibriocidal antibody titers against V. cholerae O1 Inaba and V. cholerae O1 Ogawa 4 weeks after each dose vaccination of OSP:rTTHc CCV/placebo compared to pre-vaccination.

The exploratory objectives are:

* To describe the anti tetanus toxoid (anti-TT) Immunoglobulin G (IgG) 4 weeks after each dose vaccination of OSP:rTTHc CCV/placebo compared to pre-vaccination.
* To describe memory B cell responses 4 and 28 weeks after first dose vaccination of OSP:rTTHc CCV/placebo compared to pre-vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Korean participants aged 19 to 45 years at consent
2. Participants willing to provide written informed consent to participate study voluntarily
3. Participants who can be followed up during the study period and can comply with the study requirements
4. Individual in good health as determined by the outcome of medical history, physical examination, laboratory evaluations and the clinical judgment of the investigator
5. Females of childbearing potential with negative pregnancy test result on the day of screening
6. Females of childbearing potential who agree to use an effective birth control method* from the screening and p to 12 weeks after the second dose vaccination.
7. Males who agree to use an effective birth control method* from the screening and up to 12 weeks after the second dose vaccination

Exclusion Criteria:

1. Known history or allergy to investigational vaccine components and/or excipients or other medications, or any other allergies deemed by the investigator to increase the risk of an adverse event if they were to participate in the trial
2. Individuals with major congenital abnormalities which in the opinion of investigator may affect the participant's participation in the study
3. Known history of immune function disorders including immunodeficiency diseases (known HIV infection or other immune function disorders)
4. Use of systemic steroids within past 6 months (>10 mg/day prednisone equivalent for periods exceeding 2 consecutive weeks), or receive chemotherapy, radiation therapy or other immunosuppressive drugs within the past 6 months.
5. Individuals with behavioral or cognitive impairment or psychiatric disease or neural disorders that, in the opinion of the investigator, could interfere with the participant's ability to participate in the trial
6. Individuals with splenectomy
7. Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time resulting in contraindication for intramuscular injections/blood extractions
8. Receipt of blood, blood-derived products, or immunoglobulin products in the past 3 months
9. Individuals who have received other vaccines from 4 weeks prior to the first dose of test vaccination or planned to receive any vaccine within 4 weeks of the last dose of the investigational product
10. Body mass index (BMI) ≥ 35 kg/m2
11. Individuals with active or previous Vibrio cholerae infection
12. Individuals with history of severe diarrhea requiring hospitalization or emergency room visit for the last 5 years
13. Individuals with receipt of a cholera vaccine
14. Individuals who lived in cholera endemic areas for more than 6 months for the past 10 years
15. As per Investigator's medical judgement, an individual could be excluded from the study despite meeting all inclusion/exclusion criteria mentioned above
16. Any female participant who is lactating*, pregnant or planning for pregnancy** during study period
17. Individuals enrolled in another clinical trial or bioequivalence test during 6 months prior to enrollment, concomitantly enrolled or scheduled to be enrolled in another trial
18. Individuals who are research staff involved with the clinical study or family/household members of research staff

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Serious adverse events (SAEs) and adverse events of special interest (AESIs) | Entire study participation period (approximately 7 months)
  Occurrence of any SAEs/AESIs from the time of the first dose of study vaccine
Immediate adverse events | Within 30 minutes post each dose
  Occurrence of immediate adverse events within 30 minutes from the time of each study vaccination.
Solicited adverse events | Within 7 days post each dose
  Occurrence of solicited injection site and solicited systemic adverse events from the time of each study vaccination through 7 days after each study vaccination
Unsolicited adverse events | Within 28 days post each dose
  Occurrence of unsolicited adverse events from the time of each study vaccination through 28 days after each study vaccination.
Clinical safety laboratory parameters | Within 28 days post each dose
  Occurrence of clinically significant changes in clinical safety laboratory parameters from the time of each vaccination through 28 days after each study vaccination.

SECONDARY OUTCOMES:
Seroconversion rates of IgG antibody responses to OSP | Baseline and at 28 days post the first and second dose
  Proportion of participants achieving seroconversion (defined as a 4-fold increase of serum anti-OSP IgG antibody titer at approximately 28 days after the first and second dose of investigational product compared to baseline
Geometric Mean Titers (GMTs) of serum anti-OSP IgG | Baseline and at 28 days post the first and second dose
  GMTs of serum anti-OSP IgG antibodies at 28 days after the first and second dose of investigational product compared to baseline
Geometric Mean Fold Rise (GMFR) of serum anti-OSP IgG | At 28 days post the first and second dose
  GMFR of serum anti-OSP IgG antibodies at 28 days after the first and second dose of investigational product
Seroconversion rates of serum vibriocidal antibody titers | Baseline and at 28 days post the first and second dose
  Proportion of participants with a 4-fold or greater rises in serum vibriocidal antibody titers against V. cholerae O1 Inaba and V. cholerae O1 Ogawa, relative to baseline, 28 days after the first and second dose of investigational product compared to baseline
GMT of serum vibriocidal antibody titers | Baseline and at 28 days post the first and second dose
  Geometric Mean Titers (GMT) of serum vibriocidal antibody titers against V. cholerae O1 Inaba and V. cholerae O1 Ogawa at 28 days after the first and second dose of investigational product compared to baseline
  .
GMFR of serum vibriocidal antibody titers | At 28 days post the first and second dose
  GMFR of serum vibriocidal antibody titers against V. cholerae O1 Inaba and V. cholerae O1 Ogawa at 28 days after the first and second dose of investigational product

OTHER OUTCOMES:
Seroconversion of serum anti-TT antibody titer | Baseline and at 28 days post the first and second dose
  Proportion of participants achieving seroconversion (defined as at least 4-fold increase) of serum anti-TT antibody titer at 28 days after first and second dose vaccination compared to baseline
Memory B Cell responses | Baseline, 28 days, and 6 months
  Memory B Cell responses measured by Elispot assay at 28 days after the first dose vaccination and 6 months after second dose vaccination compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Anh Wartel, MD, Principal Investigator — +82 2 8811 274
Locations (3):
- South Korea (3):
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - CHA Bundang Medical Center (CBMC) of CHA University, Seoul
  - Soon Chun Hyang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kelly M, Janardhanan J, Wagh C, Verma S, Charles RC, Leung DT, Kamruzzaman M, Pansuriya RK, Chowdhury F, Vann WF, Kaminski RW, Khan AI, Bhuiyan TR, Qadri F, Kovac P, Xu P, Ryan ET. Development of a Shigella conjugate vaccine targeting Shigella flexneri 6 that is immunogenic and provides protection against virulent challenge. Vaccine. 2024 Oct 24;42(24):126263. doi: 10.1016/j.vaccine.2024.126263. Epub 2024 Aug 31. PMID 39217775
- [Derived] Kelly M, Jeon S, Yun J, Lee B, Park M, Whang Y, Lee C, Charles RC, Bhuiyan TR, Qadri F, Kamruzzaman M, Cho S, Vann WF, Xu P, Kovac P, Ganapathy R, Lynch J, Ryan ET. Vaccination of Rabbits with a Cholera Conjugate Vaccine Comprising O-Specific Polysaccharide and a Recombinant Fragment of Tetanus Toxin Heavy Chain Induces Protective Immune Responses against Vibrio cholerae O1. Am J Trop Med Hyg. 2023 Oct 2;109(5):1122-1128. doi: 10.4269/ajtmh.23-0259. Print 2023 Nov 1. PMID 37783453